CLINICAL TRIAL: NCT06655623
Title: A Multiple Case Study of Schema Therapy for Difficult-to-treat Depression - DEPRE-ST*Case
Brief Title: A Multiple Case Study of Schema Therapy for Difficult-to-treat Depression- DEPRE-ST*Case
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Stine Bjerrum Møller, Assistant Professor, Head of Research, Region of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20220033
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Depression; Major Depressive Disorder; Chronic Depression; Treatment Resistant Depression
Keywords: schema therapy; psychotherapy; difficult-to-treat depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Schema Therapy

STUDY DESIGN:
Intervention Model Description: This study is a multiple case study of three patients with difficult-to-treat depression. The patients are also part of a larger, randomized controlled trial with two treatment arms (which also includes a Treatment As Usual arm), in which they have been assigned to the schema therapy arm.
Masking Description: The participant and investigator are both blinded to condition at the initial baseline measurements, since randomization and assignment to treatment are only made after the baseline measurements have taken place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schema therapy (Experimental): Schema therapy will be given in 30 sessions of 45-60 minutes over the course of 10-12 months. Concurrent treatment as part of the regular psychiatric treatment at the site may include psychotropic medication and 1-2 sessions with next-to-kin.
  Interventions: Behavioral: Schema therapy

INTERVENTIONS:
Behavioral: Schema therapy — Schema therapy is a form of psychotherapy invented to address more complex clinical cases. It consists of elements from Cognitive Behavioral Therapy as well as psychodynamic, emotion-focused and gestalt therapies, with a distinct focus on experiential interventions. A therapy manual was developed for use in this study.

SUMMARY:
This clinical multiple case study seeks to expand the knowledge of how schema therapy could function as an intervention for difficult-to-treat depression. The study will explore in depth the course of a 30 session treatment with schema therapy conducted over approximately one year on three individual patients at two different psychiatric treatment sites.

Together, the data from this study will inform about the feasibility of schema therapy for difficult-to-treat depression as well as form the base for recommendations in adapting schema therapy for this particular patient group.

DETAILED DESCRIPTION:
The study is part of a larger randomized controlled study, the DEPRE-ST study (clinicaltrials.gov registration: NCT05833087)(Arendt et al., 2024). The study participants will also be part of the large trial, and will be recruited for the current case study when their randomization status is being revealed; i.e., they are randomized to schema therapy.

In addition to the data collected in the DEPRE-ST trial, the patients will for each session self-report depression symptoms (before the session) and two different evaluations of the session (after the session). In addition, the patients' level of the schema therapy construct of 'Healthy Adult Mode' will be measured by self-report once monthly.

And finally, the therapist will be interviewed at the end of the treatment course about important aspects of the content and outcome of the therapy. Video recordings of each session will provide detailed information about these aspects and the interventions used in therapy.

The most important focus for the publication for this study will be to describe the trajectories of therapy for the participants, including content, effect, and subjective evaluations of therapists and participants. Also, the feasibility and adaptability of schema therapy for difficult-to-treat depression will be evaluated.

Data from outcome measurements will be presented descriptively only. Interview and video data will be compared with the outcomes measurements to reveal important events and how they might be reflected in the replies to post-session evaluation questionnaires (Session Evaluation Questionnaire and Helpful Aspects of Therapy), and in the course of the participant's self-reported depression symptoms and Healthy Adult mode.

ELIGIBILITY:
Inclusion Criteria:

* Participants have at the time of inclusion been referred to treatment for depression as a primary diagnosis in a psychiatric clinic
* Participants should meet the diagnosis of chronic or treatment-resistant depression as follows:

  1. Clinical major depression as measured by the M.I.N.I. diagnostic interview: duration minimum two years OR persistent after = 2 trials of antidepressants from different classes, in an adequate dosage and time period (= 4 weeks) OR moderate treatment resistance as measured on the MSM-scale, score > 6
  2. Minimum a score of 9 points on the Hamilton Rating Scale for Depression 6 (HAMD-6), corresponding to moderate to severe depression

Exclusion Criteria:

* Alcohol or substance abuse
* Bipolar or psychotic disorder
* Acute suicidal risk
* Mental disability (estimated IQ < 70)
* Non-Danish speaker
* Known to be pregnant at time of inclusion

Psychiatric comorbidity is not an exclusion criteria, until the comorbid disorder is understood to be the primary psychiatric problem and as such the patient would be treated in a different care package, e.g., for Post-Traumatic Stress Disorder

(The inclusion and exclusion criteria follow that of the mother study (clinicaltrial.gov ID NCT05833087))

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms, as measured with the Hamilton Depression Rating Scale 6 items (HAMD-6), self-report | Approximately once a week during the course of therapy (30-52 weeks in total), before each therapy session (30 sessions in total)
  This scale was derived from the Hamilton Depression Rating Scale 17 items and focuses on the six core symptoms of depression.

SECONDARY OUTCOMES:
Patient's experience of helpful events in therapy, as measured by the Helpful Aspects of Therapy (HAT) | Administered from the initiation of therapy, after every session (approximately once a week for 30-52 weeks, 30 sessions in total)
  The HAT was developed as a mixed qualitative and quantitative measure for describing what events in therapy were helpful or hindering for a good therapy outcome (Llewyn et al., 1988). This study will only include the first two items, which provide two blank text boxes for free writing of replies. The questions are:
  1. "Of the events which occurred in this session, which one do you feel was the most helpful or important for you personally? (By "event" we mean something that happened in the session. It might be something you said or did, or something your therapist said or did.)"
  2. "Please describe what made this event helpful/important and what you got out of it."
Patient's experiences of important aspects of the therapy session and the patient's mood in relation to the session, as measured by the Session Evaluation Questionnaire | Administered from the initiation of therapy, after every therapy session (approximately once a week, 30 sessions)
  The SEQ quantitively evaluates the psychotherapy session (9 items) and the patient's mood after the session (8 items)(the original SEQ was 21 items, but four items were removed for this study due to redundancy (Stiles et al., 1994)). Each item is scored on a bipolar, 7-point Likert scale, ranging from 1-7 and containing different, opposing aspects, e.g., 'bad-good', 'difficult-easy'. The patient is instructed to circle the appropriate number according to how they feel about the session and in themselves.
Healthy Adult schema mode, as measured on the Schema Schema Mode Inventory (SMI) - Healthy Adult subscale | Administered from the initiation of therapy - once a month, i.e. 10-12 times in total, at the end of a session of schema therapy.
  The SMI was invented to measure the psychological construct of schema modes, which are emotional activations to the activation of inherent early maladaptive schemas (cognitive constructs mostly formed in childhood)(Lobbestael et al., 2010)Reiss et al., 2016). This study will only measure the Healthy Adult mode, as the strengthening of this mode is usually an important treatment focus in schema therapy.
  The Healthy Adult mode is measured in 10 items, containing different aspects of Healthy Adult, measured on a 6 point Likert scale ranging from 'Never or almost never' to 'Always'.

OTHER OUTCOMES:
Subjective functional impairment as measured on the Work and Social Adjustment Scale (WSAS) at 6 months after baseline measurements | From baseline measurements to 6 months after baseline measurements
  5-item questionnaire
Subjective functional impairment as measured on the Work and Social Adjustment Scale (WSAS) at 12 months after baseline measurements | From baseline measurements to 12 months after baseline measurements
  5-item questionnaire
Psychological well-being as measured on the WHO-5 Well-Being Index at 6 months after baseline measurements | From baseline measurements to 6 months after baseline measurements
  5-item questionnaire
Psychological well-being as measured on the WHO-5 Well-Being Index at 12 months after baseline measurements | From baseline measurements to 12 months after baseline measurements
  5-item questionnaire
Personal recovery after mental illness as measured on the INSPIRE-O Brief at 6 months after baseline measurements | From baseline measurements to 6 months after baseline measurements
  5-item questionnaire
Personal recovery after mental illness as measured on the INSPIRE-O Brief at 12 months after baseline measurements | From baseline measurements to 12 months after baseline measurements
  5-item questionnaire
Reactions to anger as measured on the Dimensions of Anger Reactions - Revised (DAR at 6 months after baseline measurements | From baseline measurements to 6 months after baseline measurements
  7-item questionnaire
Reactions to anger as measured on the Dimensions of Anger Reactions - Revised (DAR at 12 months after baseline measurements | From baseline measurements to 12 months after baseline measurements
  7-item questionnaire
Changes in anger processing as measured on the Metacognitive Anger Processing scale Short Version (MAP) at 6 months after baseline assessments | From baseline measurements to 6 months after baseline measurements
  9-item questionnaire
Changes in anger processing as measured on the Metacognitive Anger Processing scale Short Version (MAP) at 12 months after baseline assessments | From baseline measurements to 12 months after baseline measurements
  9-item questionnaire
Changes in repetitive negative thinking as measured on the Perseverative Thinking Questionnaire (PTQ) at 6 months after baseline assessments | From baseline measurements to 6 months after baseline measurements
  15-item questionnaire
Changes in repetitive negative thinking as measured on the Perseverative Thinking Questionnaire (PTQ) at 12 months after baseline assessments | From baseline measurements to 12 months after baseline measurements
  15-item questionnaire
Negative effects of treatment as measured on the Negative Effects Questionnaire (NEQ) at 6 months after randomization | From baseline measurements to 12 months after baseline measurements
  20-item questionnaire
Negative effects of treatment as measured on the Negative Effects Questionnaire (NEQ) at 12 months after randomization | From baseline measurements to 12 months after baseline measurements
  20-item questionnaire
Changes in 1-2 patient defined problems as measured on the Psychological Outcome Profiles (PSYCHLOPS) at 6 months after baseline assessments | From baseline measurements to 6 months after baseline measurements
  Questionnaire with qualitative definition of patient defined problems and change on 6-point Likert scale
Changes in 1-2 patient defined problems as measured on the Psychological Outcome Profiles (PSYCHLOPS) at 12 months after baseline assessments | From baseline measurements to 12 months after baseline measurements
  Questionnaire with qualitative definition of patient defined problems and change on 6-point Likert scale
anxiety symptoms as measured on the Symptom Checklist-10 (SCL-10) at 6 months after baseline assessments | From baseline measurements to 6 months after baseline measurements
  5-item questionnaire - only anxiety items are used
anxiety symptoms as measured on the Symptom Checklist-10 (SCL-10) at 12 months after baseline assessments | From baseline measurements to 12 months after baseline measurements
  5-item questionnaire - only anxiety items are used
Changes in health-related quality of life as measured on the Euro-Qol-5D (EQ-5D) at 6 months after baseline assessments | From baseline measurements to 6 months after baseline measurements
  5-item questionnaire
Changes in health-related quality of life as measured on the Euro-Qol-5D (EQ-5D) at 12 months after baseline assessments | From baseline measurements to 12 months after baseline measurements
  5-item questionnaire
Prediction for treatment effect of negative expectancies for change in depression symptoms as measured on the Depression Change Expectancy Scale-pessimistic (DCES-P) items at baseline assessments | At baseline only
  11-item questionnaire - items about pessimistic expectations only
Schema modes as mediators of treatment effect after 6 months, as measured on the Schema Mode Inventory (SMI) | From baseline measurements to 6 months after baseline measurements
  37-item questionnaire - a subset of the original 118-item measure, encompassing Vulnerable Child, Healthy Adult, Demanding Critic and Punitive Critic modes
Schema modes as mediators of treatment effect after 12 months, as measured on the Schema Mode Inventory (SMI) | From baseline measurements to 12 months after baseline measurements
  118-item questionnaire
Early maladaptive schemas as measured after 6 months on the Young Schema Questionnaire 3 Short Form (YSQ-S3) | From baseline measurements to 6 months after baseline measurements
  25-item questionnaire - a subset of the original 90-item measure, encompassing the schemas Emotional Deprivation, Abandonment, Mistrust/Abuse, Social Isolation, and Defectiveness
Early maladaptive schemas as measured after 12 months on the Young Schema Questionnaire 3 Short Form (YSQ-S3) | From baseline measurements to 12 months after baseline measurements
  90-item questionnaire
Treatments for depression in earlier and current depressive episode | Collected at baseline only
  Psychotherapeutic, psychopharmacological treatment, Electroconvulsive therapy and psychiatric hospitalization, both collected from participant's given information and electronic journal records.
Childhood adversity, as measured on the Childhood Trauma Questionnaire (CTQ) | Collected at baseline only
  28-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stine B. Moeller, PhD, Principal Investigator — Region of Southern Denmark Psychiatry; University of Southern Denmark
Locations (2):
- Denmark (2):
  - Psychotherapeutic Out-patient Clinic, Psychiatric Center Copenhagen/Nannasgade, Mental Health Services, Capital Region of Denmark, Copenhagen
  - Psychotherapeutic Clinic Frederiksberg, Psychiatric Center Copenhagen, Mental Health Services, Capital Region of Denmark, Frederiksberg

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request by contacting the central contact persons of the study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available from the end of collection of data (approximately February 2026) until few years after the termination of data collection (approximately February 2031).
Access Criteria: Researchers or other professionals will gain access to all IPD upon request via a secure link/attachment provided by the study researchers.

REFERENCES:
- [Background] Arendt ITP, Gondan M, Juul S, Hastrup LH, Hjorthoj C, Bach B, Videbech P, Jorgensen MB, Moeller SB. Schema therapy versus treatment as usual for outpatients with difficult-to-treat depression: study protocol for a parallel group randomized clinical trial (DEPRE-ST). Trials. 2024 Apr 16;25(1):266. doi: 10.1186/s13063-024-08079-9. PMID 38627837
- [Background] Lobbestael J, van Vreeswijk M, Spinhoven P, Schouten E, Arntz A. Reliability and validity of the short Schema Mode Inventory (SMI). Behav Cogn Psychother. 2010 Jul;38(4):437-58. doi: 10.1017/S1352465810000226. Epub 2010 May 21. PMID 20487590
- [Background] Reiss N, Krampen D, Christoffersen P, Bach B. Reliability and validity of the Danish version of the Schema Mode Inventory (SMI). Psychol Assess. 2016 Mar;28(3):e19-26. doi: 10.1037/pas0000154. Epub 2015 Aug 10. PMID 26375430
- [Background] Llewelyn SP, Elliott R, Shapiro DA, Hardy G, Firth-Cozens J. Client perceptions of significant events in prescriptive and exploratory periods of individual therapy. Br J Clin Psychol. 1988 May;27(2):105-14. doi: 10.1111/j.2044-8260.1988.tb00758.x. PMID 3395733
- [Background] Stiles, W. B., Reynolds, S., Hardy, G. E., Rees, A., Barkham, M., & Shapiro, D. A. (1994). Evaluation and description of psychotherapy sessions by clients using the Session Evaluation Questionnaire and the Session Impacts Scale. Journal of Counseling Psychology, 41(2), 175-185. https://doi.org/10.1037/0022-0167.41.2.175